CLINICAL TRIAL: NCT04906746
Title: Pilot Study of Ruxolitinib in the Treatment of Cancer Cachexia
Brief Title: Ruxolitinib for Cancer Cachexia
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tu Dan (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor-Investigator, Tu Dan, Principal Investigator, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0475
Record Dates: First submitted 2021-05-13; First posted 2021-05-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Stage IV Non-small Cell Lung Cancer; Cachexia
Keywords: Lung cancer; Anorexia; Metabolism; Adipose; Muscle wasting
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Cachexia; Lung Neoplasms; Anorexia; Muscular Atrophy

STUDY DESIGN:
Intervention Model Description: Open label, single arm, pilot study, Intrapatient dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dosing Regimen for Ruxolitinib (Experimental): Level 0: Ruxolitinib 0 MG po bid for 1 month (Month 1)
  Level 1: Ruxolitinib 10 MG po bid for 1 month (Month 2)
  Level 2: Ruxolitinib 15 MG po bid for 1 month (Month 3)
  Interventions: Drug: Identify any dose-limiting toxicity (DLT) when ruxolitinib is administered to NSCLC cachexia patients.

INTERVENTIONS:
Drug: Identify any dose-limiting toxicity (DLT) when ruxolitinib is administered to NSCLC cachexia patients. — There will be intra-patient dose escalation of ruxolitinib in every patient enrolled on study.

SUMMARY:
To assess toxicity with use of Ruxolitinib in NSCLC cachexia patients; to associate levels of JAK/STAT signaling in blood, adipose, and muscle pre- and post-ruxolitinib treatment with changes in cachexia and anorexia.

DETAILED DESCRIPTION:
Lung cancer patients on a whole, and a significant percentage of NSCLC patients in particular, develop cancer cachexia. In fact, approximately 30-40% of all NSCLC patients will develop cachexia in their disease course, with the highest percentages in stage IV patients. One-third of these patients will die of cachexia-related morbidity. In these groups, stage-matched NSCLC patients with cachexia will have poorer survival than those without cachexia.

The JAK 1/2 inhibitor ruxolitinib has been used in many types of non-oncologic and oncologic patients with a well-established toxicity profile. Ruxolitinib was created as an oral agent with the capacity to antagonize JAK/STAT signaling across cell types. Based on the findings of the REACH2 and REACH3 trials, a starting dose of 10 mg twice daily oral administration of ruxolitinib was established for the latter patient population and is also a starting dose for the polycythemia patients. Known but manageable side effects of ruxolitinib use include thrombocytopenia, anemia, neutropenia, risk of infection, among other conditions.

Ruxolitinib has not specifically been used in 1) cancer cachexia patient populations in an evaluable trial or 2) in the setting of first line cancer therapies for solid tumors who are receiving new standards of care including immunotherapy (IO). Therefore, in this trial, investigators propose using ruxolitinib in an open-label approach to antagonize systemic and tissue-specific, tumor-directed JAK/STAT signaling as a means curtailing cachexia progression in stage IV NSCLC patients. This study will ensure an acceptable toxicity profile when ruxolitinib is used in cancer cachexia patients.The use of ruxolitinib dose escalation in the same patients with frequent tissue and serum collections will permit us to better understand how important JAK/STAT signaling is to clinical cancer cachexia development.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects at least 18 years of age;
2. Ability to understand and the willingness to sign a written informed consent;
3. Histological or biopsy proven Non-Small Cell Lung Cancer (squamous or non-squamous);
4. ECOG performance status of 0-2;
5. Patients with evidence of:

   * cancer cachexia, defined by the International Cancer Cachexia Consensus Definition (>5% weight loss over the preceding 6 months prior to diagnosis); OR
   * Patients with evidence of cancer pre-cachexia, defined by the International Cancer Cachexia Consensus Definition (0 to <=5% weight loss over the preceding 6 months prior to diagnosis);
6. Any de novo stage IV NSCLC disease diagnosis as defined by AJCC 8th edition staging. Staged with PET/CT, MRI brain, or other acceptable staging tool; measurable disease as defined by RECIST 1.1;
7. Adequate end-organ function, based on routine clinical and laboratory workup and institutional guidelines, as determined by oncology team offering patient standard of care therapy, including:

   1. ANC >1,000 cells/µl, Platelets > 100,000 cells/µl, Hemoglobin > 10.0 g/dl;
   2. Serum creatinine ≤ 1.5 x ULN or calculated creatinine clearance ≥ 45 ml/min;
   3. Total bilirubin ≤ 1.5 x ULN (or direct bilirubin below the ULN), AST and ALT ≤ 2.5 x ULN;
   4. International normalized ratio (INR) (or prothrombin time (PT)) and activated partial thromboplastin time (aPTT) ≤ 1.5 x ULN unless participant is receiving anticoagulant therapy, if values are within the intended therapeutic range;
8. Women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately; A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: a. Has not undergone a hysterectomy or bilateral oophorectomy; or b. Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months);
9. Male subjects who are surgically sterile or are using a medically acceptable form of contraception for 90 days following the completion of therapy;
10. Life expectancy anticipated to be 6 months or greater;
11. No prior therapy for advanced lung cancer.

Exclusion Criteria:

1. Subjects with confirmed stage I-III NSCLC;
2. Patients whose tumors have actionable mutations treatable with targeted therapies;
3. Patients with no evidence of cancer cachexia, defined by the International Cancer Cachexia Consensus Definition (>5% weight loss over the preceding 6 months prior to diagnosis); OR Patients with no evidence of cancer pre-cachexia, defined by the International Cancer Cachexia Consensus Definition (0 to <=5% weight loss over the preceding 6 months prior to diagnosis);
4. Active malignancy other than lung cancer that requires concurrent treatment other than hormonal therapy and is deemed by the treating physicians to be likely to affect the subject's survival duration;
5. Subjects who have not recovered or have disease control from prior treatment-related to toxicities judged by treating physician;
6. History of allergic reactions attributed to compounds of similar chemical or biologic composition to ruxolitinib or other agents used in study;
7. Uncontrolled intercurrent illness including, but not limited to, serious ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements;
8. Inadequate liver or renal function, if out of the acceptable ranges of the inclusion criteria;
9. Significant bacterial, fungal, parasitic, or viral infection requiring treatment;
10. Previous treatment with a JAK inhibitor;
11. Uncontrolled congestive heart failure (New York Heart Association Classification 3 or 4), angina, myocardial infarction, cerebrovascular accident, coronary/peripheral artery bypass graft surgery, transient ischemic attack, or pulmonary embolism within 3 months prior to initiation of ruxolitinib;
12. Females who are pregnant, breast-feeding or plan to become pregnant;
13. Participation in other clinical trials either to treat diagnosed lung or other cancers (patients on registry trials are eligible);
14. Requirement for treatment with drugs that may, in the judgment of the treating investigator, create a risk for a precipitous change in patient's health;
15. Any other conditions that, in the Investigator's opinion, might indicate the subject to be unsuitable for the study;
16. Life expectancy of less than 6 months;
17. Prior therapy for the newly diagnosed advanced lung cancer.
18. Patients taking therapies that are strong CYP3A4 inhibitors and fluconazole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2024-09-27 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of non-small cell lung cancer cachexia patients with toxicity with the use of Ruxolitinib | 3 months
  To assess toxicity with use of Ruxolitinib in NSCLC (non-small cell lung cancer) cachexia patients; to associate levels of JAK/STAT (Janus kinase-signal transducer and activator of transcription) signaling in blood, adipose, and muscle pre- and post-ruxolitinib treatment with changes in cachexia and anorexia. NCI's CTCAE v5.0 toxicity criteria will be used to measure Ruxolitinib-related side effects. Immunoblotting, FACS analyses, and other biologic metrics will be used to determine if Ruxolitinib can suppress cachexia-associated JAK/STAT activation in blood and peripheral tissues.

SECONDARY OUTCOMES:
Number of adverse events associated with ruxolitinib when administered to cancer cachexia patients | 3 months
  For the secondary objective of adverse events, investigator will again use NCI's CTCAE v5.0 toxicity criteria throughout the trial evaluation.
Number of participants with Objective Response (OR) as determined by RECIST criteria | 3 months
  Patient tumor response will be determined by CT-based imaging (CT, PET/CT), MRI (brain evaluation), and other clinical indicators (bronchoscopy, image-guided biopsies), etc. with RECIST and iRECIST criteria response criteria as a function of Ruxolitinib use and dose. In patients with measurable disease, to describe any preliminary evidence of Ruxolitinib's anti-tumor activity by assessment of objective response as determined by RECIST in cancer cachexia patients. Two such measurements will be conducted during the course of the trial.
Analysis providing any preliminary evidence that ruxolitinib improves quality of life (QoL) for cancer cachexia patients | 4 months
  Quality of life questionnaire while on ruxolitinib will be assessed with the EORTC QLQ-CAX24 (The European Organization for Research and Treatment of Cancer quality of life questionnaire). Questionnaire will be given to patients every 2 weeks for 3 months while on study and 1 month of follow-up.
Suppression of body weight loss in cancer cachexia patients | 4 months
  To describe any preliminary evidence suggesting that Ruxolitinib suppresses body weight loss in cancer cachexia patients. Body weight will be measured every 2 weeks while on study, including 1 month of follow-up, to provide measures of how Ruxolitinib may be suppressing cachexia-associated body weight loss.
Analysis of any preliminary evidence suggesting that Ruxolitinib suppresses adipose and lean muscle loss in cancer cachexia patients. | 4 months
  Body weight will be measured every 2 weeks while on study, including 1 month of follow-up. Both DEXA (dual-energy x-ray absorptiometry) imaging every 2 weeks while on study/follow-up and CT-based imaging with auto-segmentation will provide measures of how Ruxolitinib may be suppressing cachexia-associated adipose and muscle loss.
Analysis of any preliminary evidence suggesting that Ruxolitinib suppresses anorexia in cancer cachexia patients. | 4 months
  Anorexia will be assessed with the EORTC QLQ-CAX24 questionnaire as well as direct clinical history taking every 2 weeks on study. Descriptive statistics will be used to report changes.
Analysis of any preliminary evidence suggesting that Ruxolitinib improves overall survival in cancer cachexia patients. | 6 months
  Progression-free survival (CT-based imaging) will be assessed for all patients while on and off Ruxolitinib. There will be one determination of OS at 6 months from start of active phase of study. Estimates will be descriptively presented using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Tu Dan, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States